CLINICAL TRIAL: NCT06580288
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Finerenone in the Treatment of IgA Nephropathy
Brief Title: Effect of Finerenone in IgA Nephropathy
Acronym: FIGHT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Du Xiaoying, chief physician, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20240069C-R1
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finerenone (Experimental)
  Interventions: Drug: Finerenone
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone — 10mg or 20mg
  Arms: Finerenone
Drug: Placebo — 10mg or 20mg
  Arms: placebo

SUMMARY:
The aim of this trial is to conduct a randomized, multicenter, placebo-controlled, double-blind clinical trial to determine the safety and efficacy of Finerenone in reducing proteinuria and protecting renal function in patients with IgA nephropathy.

The primary endpoint event was the change in urinary albumin/creatinine ratio between the two groups at 12 months of treatment.

DETAILED DESCRIPTION:
This is a randomized, multicenter, placebo-controlled, double-blind clinical trial aimed at clarifying the safety and efficacy of finerenone in reducing proteinuria and protecting renal function in patients with IgA nephropathy.

Study population will include participants with renal biopsy confirmed IgA nephropathy (eGFR ≥ 30 mL/min/1.73 m2) and UACR ≥500mg/g ≤3500mg/g. Participants receiving maximum tolerated dose of RAS inhibitor treatment for more than 3 months are eligible for the study.

The study will be conducted at 4 sites. 120 participants will be randomised to one of 2 arms in a 1:1 ratio:

* Finerenone 10mg/20 mg
* Placebo 10mg/20 mg For each participant, the total duration of participation will be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Kidney biopsy confirmed IgA nephropathy within 2 years, with secondary IgA nephropathy excluded;
* Age ≥ 18 years;
* Maximum tolerated dose of RAS inhibitors for more than 3 months, with urine albumin/creatinine ratio ≥ 500 mg/g and ≤ 3500 mg/g; V1 laboratory test showing urine albumin/creatinine ratio ≥ 500 mg/g and ≤ 3500 mg/g. After maximum tolerated dose of RAS inhibitors or ARB, V2 urine albumin/creatinine ratio ≥ 500 mg/g and ≤ 3500 mg/g;
* eGFR calculated by EPI ≥ 30 ml/min/1.73 m²;
* Serum potassium level ≤ 4.8 mmol/L;
* SBP ≤ 150 mmHg, DBP ≤ 110 mmHg;
* LVEF > 40%;
* Willing and able to provide informed consent.

Exclusion Criteria:

* There are clear indications for the use of immunosuppressive therapy, such as: nephrotic syndrome (urine protein greater than 3.5 g/d, blood albumin less than 30 g/L), pathological minimal change disease combined with IgA nephropathy; the proportion of crescents in kidney biopsy is ≥ 50%.
* Any existing life-threatening condition with a life expectancy of less than 2 years;
* Active infection, HBV infection, or active lesions (nodules, cavities, or tuberculomas);
* AKI causing renal dysfunction;
* Use of steroids/immunosuppressive drugs within the past 3 months;
* History of malignant tumors, regardless of treatment status or evidence of local recurrence or metastasis;
* Any surgical or medical condition that may significantly alter the absorption, distribution, metabolism, or excretion of the investigational drug;
* History of drug or alcohol abuse within the past 12 months;
* History of drug allergies or contraindications;
* Previous noncompliance or unwillingness to follow the study protocol;
* Any condition that may affect safety or efficacy;
* History of kidney transplantation or currently receiving immunosuppressive treatment;
* Pregnant or breastfeeding women;
* Obese patients with a BMI > 35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
change in uACR between the two groups | at 12months

SECONDARY OUTCOMES:
eGFR slop | at 12months
change in uPCR between the two groups | at 12months
renal failure (eGFR decline of 40% or progression to ESKD, defined as initiation of dialysis, kidney transplantation, or eGFR ≤ 15 ml/min/1.73 m²); | at 12months
cardiovascular event endpoints: cardiovascular death or non-fatal myocardial infarction or non-fatal stroke; hospitalization due to heart failure; major cardiovascular events; all-cause mortality. | at 12months

IPD SHARING:
Plan to Share IPD: No